CLINICAL TRIAL: NCT00239252
Title: Comparison in Efficacy and Safety Between Interferon Alfacon-1 Alone and Concomitant Dosing With Ribavirin for the Treatment of Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B6431/HCT1
Record Dates: First submitted 2005-09-13; First posted 2005-10-17 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C
Keywords: Interferon alfacon-1; Virus disease; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Virus Diseases | interventions — interferon alfacon-1

INTERVENTIONS:
Drug: Interferon alfacon-1

SUMMARY:
Efficacy and safety is compared between interferon alfacon-1 alone and concomitant dosing of interferon alfacon-1 and ribavirin in hepatitis C patients.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C patients (high titer, genotype1)

Exclusion Criteria:

* Patients with autoimmune disorder
* Patients with negative HBs antigen
* Patients with hepatic cirrhosis, hepatic failure and hepatic cancer
* Patients with depression or psychoneurotic disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development III, Study Chair — Astellas Pharm. Inc.
Locations (5):
- Japan (5):
  - Chubu Region
  - Chugoku Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region